CLINICAL TRIAL: NCT05546346
Title: Clinical Application of Wearable Magnet Tracking System for Capsule Endoscopes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2022SDU-QILU-827
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Capsule Endoscopes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- wearable magnet tracking system (Experimental)
  Interventions: Device: wearable magnet tracking system

INTERVENTIONS:
Device: wearable magnet tracking system — In this group, wearable magnet tracking system was used.

SUMMARY:
The investigators developed a wearable magnet tracking system, which provided a non-invasive and high accuracy method for capsule endoscopes localization. Data fusion from multiple sensors expanded positioning range and proposed localization algorithm overcame shortcomings of existing systems. This clinical trial was conducted to verify effectiveness and stability of the tracking system.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 75
* agree to give written informed consent

Exclusion Criteria:

* dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis, overt gastrointestinal bleeding, history of upper gastrointestinal surgery or abdominal surgery altering gastrointestinal anatomy, or postabdominal radiation
* congestive heart failure, renal insufficiency, under therapeutic anticoagulation, in poor general condition (American Society of Anesthesiologists class III/IV), claustrophobia, metallic parts, a pacemaker or other implanted electromedical devices, or artificial heart valves
* pregnancy or suspected pregnancy
* exclusion criteria for standard magnetic resonance imaging examination such as the presence of surgical metallic devices, even though its low magnetic field technically would not interferewith such devices
* currently participating in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The duration of time | 12 months
  the length of time of the tracking system used in continuous acquisition of the magnetic field strength values

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China